CLINICAL TRIAL: NCT04663217
Title: Exercise Hemodynamic, Right Ventricular Coupling and Echocardiography in Pulmonary Hypertension
Acronym: EXERTION
Status: Completed | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Other Study IDs: AZ 11716
Record Dates: First submitted 2020-11-05; First posted 2020-12-10 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Hypertension, Pulmonary; Hypertension, Pulmonary Arterial
Keywords: exercise; Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pulmonary arterial hypertension: Patients with mean pulmonary arterial pressure above 25 mmHg, and a pulmonary capillary wedge pressure below 15 mmHg classified into group 1 of the clinical classification of pulmonary hypertension.
  Interventions: Other: Exercise
- Pulmonary hypertension due to left heart disease: Patients with mean pulmonary arterial pressure above 25 mmHg, and a pulmonary capillary wedge pressure above 15 mmHg with left heart disease, classified into group 2 of the clinical classification of pulmonary hypertension.
  Interventions: Other: Exercise
- Chronic thromboembolic pulmonary hypertension: Patients with mean pulmonary arterial pressure above 25 mmHg, and a pulmonary capillary wedge pressure below 15 mmHg with a history of pulmonary embolism, classified into group 4 of the clinical classification of pulmonary hypertension.
  Interventions: Other: Exercise
- Control: Patients with mean pulmonary arterial pressure below 25 mmHg, and a pulmonary capillary wedge pressure below 15 mmHg with exclusion of pulmonary hypertension.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — After placement of the right heart catheter patients will undergo an exercise challenge in semi-supine position until exhaustion

SUMMARY:
This study aims to investigate the exercise profile in pulmonary hypertension patients with either pulmonary arterial hypertension, chronic thromboembolic pulmonary hypertension or pulmonary hypertension due to left heart disease and in disease control.

DETAILED DESCRIPTION:
This is a dual-center observational prospective study in patients with pulmonary arterial hypertension, chronic thromboembolic pulmonary hypertension, pulmonary hypertension due to left heart disease. Patients undergoing right heart catheterisation due to dyspnoe with invasive exclusion of pulmonary hypertension will be recruited as disease control.

The study comprises a 1-day screening period, followed by a right heart catheterization with exercise challenge.

The study starts with screening, information of the patients and Informed Consent Form signature at day -1. Screening and inclusion of the patient can be performed on the same day. On the day of the planned right heart catheterization based on clinical grounds, exercise right heart catheterisation (RHC) using Swan-Ganz and/or Conductance catheters with simultaneous echocardiography will be performed. End of study is defined as a complete exercise RHC. Adverse events will be assessed until 1 day after the exercise RHC.

After placement of the Swan-ganz or Conductance catheter patients will undergo an exercise challenge using the following protocol in semi-supine position until exhaustion:

* Incremental workload increase of 20Watt every 2-4 min.
* For patients not able to start a 20 Watt, initial workload can be adjusted to a minimum of 5 Watt with 5 Watt increase every 2-4 min until exhaustion
* Maximal exercise duration is 10-12 minutes
* Symptoms of dyspnoea during exercise will be rated by subjects at baseline, after 6 minutes and at maximum according to the Borg perceived dyspnoea (0-10) scale.

Simultaneously, echocardiography and lung ultrasound will be performed before exercise (baseline), after 6 minutes of exercise and at maximum.

After assessment of right ventriclure pressure-volume loops during maximum exercise, guided by echocardiographic the conductance catheter will be placed in the right atrium to obtain right atrium pressure-volume loops during maximum exercise.

Optional, the exercise RHC will be performed without the Conductance catheter and only with the Swan-Ganz catheter. In this case, pressure values and cardiac output will be measured using the thermodilution method, averaging 3-5 measurements at baseline, 6 minutes and maximum. Detailed assessment of right atrial pressure curves (with a and v wave) will be performed at baseline, 6 minutes and maximum exercise.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of pulmonary arterial hypertension (World Health Organization group 1)
* Pulmonary hypertension due to left heart disease (World Health Organization group 2)
* Chronic thromboembolic pulmonary hypertension (World Health Organization group 4)
* Invasive exclusion of pulmonary hypertension
* Age ≥ 18 years
* Planned right heart catheterization based on clinical grounds
* Stable specific PAH medications
* Ability to undergo cycle ergometry
* Signed informed consent

Exclusion Criteria:

* Other etiologic groups of pulmonary hypertension (World Health Organization group 3, 5)
* Unstable or severe coronary artery disease
* Uncontrolled arterial hypertension
* Left ventricular ejection fraction < 30%
* Severe congenital or acquired valvular or myocardial disease
* Progressive left heart failure
* History of severe ventricular arrhythmias
* Severe, terminal renal impairment
* Severe obstructive or restrictive lung disease
* Severe lung emphysema or interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Confirmed diagnosis of either pulmonary arterial hypertension; pulmonary hypertension due to left heat disease; chronic thromboembolic pulmonary hypertension; or invasive exclusion of pulmonary hypertension (control group)
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2023-11-04 (Actual)

PRIMARY OUTCOMES:
exercise pulmonary arterial pressure | 1 day
  mean pulmonary arterial pressure (mmHg)
exercise cardiac output | 1 day
  cardiac output (l/min);
exercise pulmonary wedge pressure | 1 day
  pulmonary arterial wedge pressure (mmHg)
exercise arterial elastance | 1 day
  arterial elastance (mmHg/mL)
exercise end-systolic elastance | 1 day
  end-systolic elastance (mmHg/mL)
exercise mean right atrial pressure | 1 day
  mean right atrial pressure (mmHg)
exercise right atrial function | 1 day
  right atrial strain (%)
exercise right volume | 1 day
  right ventricular volume (ml)
exercise right ventriculare function | 1 day
  right ventricular strain (%)
exercise right atrial volume-pressure curves | 1 day
  atrial volume to pressure ratio (ml/mmHg)

SECONDARY OUTCOMES:
exercise lung congestion | 1 day
  B-Lines
exercise left atrial function | 1 day
  left atrial strain (%)
exercise left atrial volume | 1 day
  left atrial volume (ml)
exercise hepatic backflow | 1 day
  diameter inferior vena cava (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Richter J Manuel, MD, Principal Investigator — UKGM Giessen
Locations (2):
- Germany (2):
  - Kerckhoff-Klinik, Bad Nauheim, Hesse
  - University of Giessen, Giessen, Hesse

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon request.

REFERENCES:
- [Derived] Yogeswaran A, da Rocha BB, Rako ZA, Kaufmann SJ, Schafer S, Kremer N, Ghofrani HA, Seeger W, Tello K. Physiological mechanisms behind respiratory variations in right atrial pressure in pulmonary hypertension. Sci Rep. 2024 May 31;14(1):12547. doi: 10.1038/s41598-024-61825-6. PMID 38822042
- [Derived] Rako ZA, Yogeswaran A, Lakatos BK, Fabian A, Yildiz S, da Rocha BB, Vadasz I, Ghofrani HA, Seeger W, Gall H, Kremer NC, Richter MJ, Bauer P, Tedford RJ, Naeije R, Kovacs A, Tello K. Clinical and functional relevance of right ventricular contraction patterns in pulmonary hypertension. J Heart Lung Transplant. 2023 Nov;42(11):1518-1528. doi: 10.1016/j.healun.2023.07.004. Epub 2023 Jul 13. PMID 37451352